CLINICAL TRIAL: NCT03250598
Title: A Phase 1, Single-Dose, Open-Label Study to Characterize and Compare the Pharmacokinetics, Safety, and Effect on QTc Interval of AG-348 in Healthy Subjects of Japanese Origin and Healthy Subjects of Non-Asian Origin
Brief Title: Study to Evaluate the Pharmacokinetics, Safety, and QTc Effect of AG-348 in Healthy Subjects of Japanese Origin and Non-Asian Origin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: AG348-C-004
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Healthy; Japanese; Non-Asian
Keywords: Healthy; Japanese
MeSH Terms: interventions — mitapivat

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental)
  Interventions: Drug: AG-348
- Cohort B (Experimental)
  Interventions: Drug: AG-348
- Cohort C (Experimental)
  Interventions: Drug: AG-348

INTERVENTIONS:
Drug: AG-348 — 50 mg single-dose
  Arms: Cohort A
Drug: AG-348 — 5 mg single-dose
  Arms: Cohort B
Drug: AG-348 — 200 mg single-dose
  Arms: Cohort C

SUMMARY:
The purpose of this Phase I, single-dose, open-label trial is to evaluate the pharmacokinetics, safety, and effect on QTc interval of AG-348 in healthy, adult Japanese and Non-Asian subjects. The study plans to evaluate 3 cohorts of a single oral dose of AG-348 in Japanese and Non-Asian subjects. Pharmacokinetic sampling will take place serially at specified times during conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

* Be a male or female aged 18 to 55 years, inclusive.
* Have a body mass index (BMI) of ≥ 18.5 to ≤ 29.0 kg/m2 at Screening.
* Be healthy overall with no clinically significant medical abnormalities, as determined by the Investigator through evaluation of the subject's medical history and Screening vital signs, ECG, physical examination, and laboratory assessments.
* Applicable to Japanese Subjects Only: Japanese subjects must have been born in Japan, have both parents and all grandparents of Japanese origin, and not have lived outside of Japan for more than 5 years with no significant changes in lifestyle, including diet, since leaving Japan.
* Applicable to Non-Asian Subjects Only: Non-Asian subjects must have both parents and all grandparents of Non-Asian origin.

Exclusion Criteria:

* Have undergone any major surgical procedure within the 3 months prior to Screening.
* Test positive at Screening for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), or human immunodeficiency virus (HIV).
* Have a Screening systolic blood pressure (BP) reading of > 140 mmHg (> 150 mmHg in subjects > 45 years of age) OR a diastolic BP reading of > 90 mmHg after 5 minutes of supine rest.
* Have any of the following cardiac risk factors:

  1. Be taking any medication with a known effect of QT interval prolongation (see list of medications in Appendix 1)
  2. Have a cardiac pacemaker
  3. Demonstrate on either the Screening ECG or the baseline ECG any evidence of atrial fibrillation, atrial flutter, complete right or left bundle branch block, or Wolff-Parkinson-White syndrome
  4. Demonstrate on the Screening ECG any morphology that renders measurement of QT interval imprecise (eg, neuromuscular artifact that cannot be readily eliminated, indistinct QRS onset, low-amplitude T wave, merged T and U waves, prominent U waves, arrhythmia)
* Have a history of a known risk factor for Torsade de Pointes, including any of the following:

  1. Personal or family history of congenital long QT syndrome, Brugada syndrome, or sudden death
  2. Unexplained syncope
  3. Heart failure
  4. Myocardial infarction
  5. Angina
  6. Certain clinically significant laboratory assessment findings, including hypokalemia, hypercalcemia, or hypomagnesemia
* Have had, including by voluntary donation, > 400 mL of blood collected within the 3 months prior to Screening.
* Have taken within the 14 days prior to study drug dosing any prescription medication, over-the counter medication, or nonprescription preparation-including vitamins, minerals, phytotherapeutic/herbal/plant-derived preparations, or grapefruit juice-unless deemed acceptable by the Investigator OR have taken within the 28 days prior to study drug dosing any restricted product known to strongly induce CYP3A4 metabolism (eg, St. John's Wort).
* Have participated in another clinical research study within the 3 months prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2017-10-09 (Actual)

PRIMARY OUTCOMES:
AUC | Pharmacokinetic sampling for AG-348 will be taken for 72 hours (4 days) after single dose
  AG-348 Area Under the Curve
Cmax | Pharmacokinetic sampling for AG-348 will be taken for 72 hours (4 days) after single dose
  AG-348 Maximum Plasma Concentration

SECONDARY OUTCOMES:
Incidence of Adverse Events | 10 (± 1) days after single-dose of AG-348
  Assessment of adverse events
QTc interval | Change in QTc from baseline will be presented by race and by cohort
  QTc interval measurements

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs Agios Pharmaceuticals, Inc, Study Chair — Agios Pharmaceuticals, Inc.
Locations (1):
- West Coast Clinical Trial (WCCT) Global, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No